CLINICAL TRIAL: NCT02053272
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Group, Dose Ranging Study of GWP42004 as Add on to Metformin in the Treatment of Participants With Type 2 Diabetes
Brief Title: A Study of GWP42004 as Add on to Metformin in the Treatment of Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWDM1302; 2013-001140-61 (EudraCT Number)
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Glycaemic control; Delta-9-tetrahydrocannabivarin; Cannabinoids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 mg GWP42004 bid (Active Comparator): Licaps® size double zero (Size 00) hard gelatin capsules containing 2 mg GWP42004 dissolved in excipients Macrogolglycerol Ricinoleate and Oleoyl macrogol-6-glycerides. One capsule taken twice daily for 12 weeks.
  Interventions: Drug: GWP42004
- 5 mg GWP42004 bid (Active Comparator): Licaps® size double zero (Size 00) hard gelatin capsules containing 5 mg GWP42004 dissolved in excipients Macrogolglycerol Ricinoleate and Oleoyl macrogol-6-glycerides. One capsule taken twice daily for 12 weeks.
  Interventions: Drug: GWP42004
- 15 mg GWP42004 bid (Active Comparator): Licaps® size double zero (Size 00) hard gelatin capsules containing 15 mg GWP42004 dissolved in excipients Macrogolglycerol Ricinoleate and Oleoyl macrogol-6-glycerides. One capsule taken twice daily for 12 weeks.
  Interventions: Drug: GWP42004
- Placebo (Placebo Comparator): Licaps® size double zero (Size 00) hard gelatin capsules containing excipients Macrogolglycerol Ricinoleate and Oleoyl macrogol-6-glycerides. One capsule taken twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42004 — The total dose administered within any 24-hour interval will be two capsules (typically 12 hours apart).
  Other Names: Delta-9-tetrahydrocannabivarin
  Arms: 15 mg GWP42004 bid; 2 mg GWP42004 bid; 5 mg GWP42004 bid
Drug: Placebo — The total dose administered within any 24-hour interval will be two capsules (typically 12 hours apart).
  Other Names: Placebo control
  Arms: Placebo

SUMMARY:
A study to compare the change in glycaemic control in participants with Type 2 diabetes when treated with GWP42004 or placebo as add-on therapy to metformin over a period of 12 weeks. The safety and tolerability of GWP42004 compared with placebo will also be assessed.

DETAILED DESCRIPTION:
This 14 week (one week baseline, 12 week treatment period and one week follow-up), multicentre, randomised, double blind, placebo controlled, parallel group study will evaluate the efficacy, safety and tolerability of 2, 5 and 15 mg of GWP42004 as add on to metformin compared with placebo in participants with Type 2 diabetes.

Eligible participants will enter the study at a screening visit (Visit 1, Day -7) where the following information will be obtained for each participant:

1. Informed consent
2. Demographics
3. Medical history
4. Concomitant medications
5. Electrocardiogram (ECG)
6. Physical examination
7. Vital signs
8. Body weight
9. Height
10. Body Mass Index (BMI)
11. Beck Depression Inventory-II (BDI-II)
12. Safety blood test (biochemistry and haematology)
13. Efficacy blood test (HbA1c)
14. Urinalysis (including drugs of abuse screen)
15. Pregnancy test (if appropriate)

Once all inclusion and exclusion criteria have been reviewed, participants will be commence a seven day baseline period. The day before Visit 2, participants will perform blood glucose tests and record the results, along with the associated time of assessment, in the study diary. Participants will then fast overnight.

Participants will return to the clinic at Visit 2 (Day 1) and following review of all inclusion and exclusion criteria, the following information will be obtained for each participant:

1. Body weight
2. BMI
3. Physical examination
4. Vital signs
5. Safety blood test (biochemistry and haematology)
6. GWP42004 exposure blood test (plasma levels)
7. Efficacy blood test (HbA1c, fasting plasma glucose, serum fructosamine, fasting plasma insulin, HOMA2-IR, pro-insulin, C-peptide, HOMA2-%B, total cholesterol, HDL-cholesterol, serum triglycerides, C-reactive protein)
8. Urinalysis
9. Concomitant medications
10. Adverse events (AEs)
11. BDI-II
12. Columbia-Suicide Severity Rating Scale (C-SSRS)
13. Diabetes Treatment Satisfaction Questionnaire (DTSQs)
14. Overall health Visual Analogue Scale (VAS)
15. Cannabis withdrawal scale assessment (UK only).

Participants will then be randomised to receive either GWP42004 (2, 5 or 15 mg bid) or placebo to be taken adjunctive to their currently prescribed medication. The first dose will be administered and a Oral Glucose Tolerance Test (OGTT) performed.

A third (Visit 3, Day 29) and fourth (Visit 4, Day 57) visit will take place mid-treatment. The day before these visits, participants will perform blood glucose tests and record the results, along with the associated time of assessment, in the study diary. Participants will then fast overnight. The following information will be obtained for each participant at Visits 3 and 4:

1. Body weight
2. BMI
3. Physical examination
4. Vital signs
5. Safety blood test (biochemistry and haematology)
6. Efficacy blood test (HbA1c, fasting plasma glucose, fasting plasma insulin, HOMA2-IR, HOMA2-%B)
7. Urinalysis
8. Concomitant medications
9. AEs
10. BDI-II
11. C-SSRS
12. DTSQs
13. Overall health VAS

A cannabis withdrawal scale assessment will be made by telephone (UK only) between Visits 4 and 5.

A further visit will take place at the end of treatment (Visit 5, Day 85). Two days before this visit, a cannabis withdrawal scale assessment will be made by telephone (UK only). The day before Visit 5, participants will perform blood glucose tests and record the results, along with the associated time of assessment, in the study diary. Participants will then fast overnight. The following information will be obtained for each participant at Visit 5:

the following information will be obtained for each participant:

1. Body weight
2. BMI
3. Physical examination
4. ECG
5. Vital signs
6. Safety blood test (biochemistry and haematology)
7. GWP42004 exposure blood test (plasma levels)
8. Efficacy blood test (HbA1c, fasting plasma glucose, serum fructosamine, fasting plasma insulin, HOMA2-IR, pro-insulin, C-peptide, HOMA2-%B, total cholesterol, HDL-cholesterol, serum triglycerides, C-reactive protein)
9. Urinalysis (including drugs of abuse screen)
10. Pregnancy test (if appropriate)
11. Concomitant medications
12. Adverse events (AEs)
13. BDI-II
14. OGTT
15. C-SSRS
16. DTSQs
17. Overall health VAS

One, three and seven days following Visit 5 (Days 86, 89 and 92, respectively), further cannabis withdrawal scale assessments will be made by telephone (UK only). A final review of AEs and concomitant medications will be made by telephone to all participants on Day 92.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study (see Section 15.2).
* Male or female participants aged 18 years or above.
* Clinically diagnosed with Type 2 diabetes.
* Participants receiving oral metformin (≥1000 mg per day) as anti-diabetic treatment who have received a stable dose for at least three months prior to enrolment (Visit 1) and willing to maintain a stable dose for the duration of the trial.
* HbA1c level of >7% - ≤9% (53 - 74.9 mmol/mol).
* BMI of >25 - <40 (>23 - <40 for Asian populations).
* No changes in diet or exercise for three months prior to study entry and participant agrees to keep stable for the duration of the study.
* Capable of complying with the study requirements and completing the study (in the opinion of the investigator).
* Participant is able (in the investigators opinion) and willing to comply with all study requirements.
* Participant is willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Participant is willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Participant is taking or has taken insulin at any point in the last year (does not include short term use (<10 days) to treat acute events).
* Participant is taking or has taken anti-diabetic treatment (other than metformin) in the three months prior to screening.
* Any concomitant medications which, in the opinion of the investigator, could affect the primary endpoint should remain stable or not be prescribed in the one month prior to Visit 1 or during the study period.
* Any known of suspected history of:
* Alcohol or substance abuse.
* Epilepsy or recurrent seizures.
* Participants receiving treatment with antidepressants or under observation for depression.
* BDI-II item 9 score of 1, 2 or 3.
* Participant who has significant history of suicidal ideation or self-harm.
* Recent (within three months of screening) blood loss (including blood donation).
* Haemolytic anaemia.
* Genetic abnormality in haemoglobin molecule (e.g. sickle cell anaemia).
* Clinically significant cardiac, renal or hepatic impairment in the opinion of the investigator.
* Has significantly impaired renal function as evidenced by a creatinine clearance lower than 40 mL/min at Visit 1.
* Has significantly impaired hepatic function at Visit 1 (alanine aminotransferase (ALT) levels >5x upper limit of normal (ULN) or total bilirubin (TBL) levels > 2x ULN). If the ALT or aspartate aminotransferase (AST) levels are >3x ULN and the TBL levels >2x ULN (or International Normalised Ratio (INR) >1.5), then this participant should not enter the study.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMPs.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective double barrier contraception.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Participants who have received an Investigational Medicinal Product (IMP) within the 12 weeks prior to the screening visit.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, may influence the result of the study, or the participant's ability to participate in the study.
* Following a physical examination, the participant has any abnormalities that, in the opinion of the investigator would prevent the participant from safe participation in the study.
* Unwilling to abstain from donation of blood during the study.
* Participants who have previously undergone bariatric surgery.
* Travel outside the country of residence planned during the study, unless the participant has prior permission from the embassy of the destination country.
* Participants previously randomised into this study.
* The patient is currently using or has used cannabis or cannabinoid based medications within 30 days of study entry and is unwilling to abstain for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of treatment in mean glycosylated haemoglobin A1c (HbA1c) level. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of HbA1c levels. Values are calculated as a percentage of total haemoglobin. A decrease from baseline to the end of treatment in base per cent values, a negative value, indicates an improvement.

SECONDARY OUTCOMES:
Change from baseline to the end of treatment in mean fasting plasma glucose concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of fasting plasma glucose concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean serum glucose concentration two hours post glucose challenge (Oral Glucose Tolerance Test [OGTT]) | Baseline (Day 1) and End of treatment (Day 85)
  Fasting blood samples are taken at 0 minutes prior to a glucose drink and at 30 and 120 minutes post drink. The OGTT measures the serum glucose levels at two hours (120 minutes) compared to 0 minutes. The extent of the elevation in serum glucose levels following a glucose drink are compared between baseline and the end of treatment. A reduction in the elevation of serum glucose levels at the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean serum fructosamine concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of serum fructosamine concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in the number of participants with a HbA1c level below 7%. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of glycosylated haemoglobin A1c levels. Values are calculated as a percentage of total haemoglobin. An increase in the number of participants with HbA1c levels below 7% from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean fasting plasma insulin concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of fasting plasma insulin concentrations. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean insulin resistance measured by Homeostasis Model Assessment 2 (HOMA2-IR). | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of insulin resistance calculated by HOMA2-IR. HOMA2-IR is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin resistance, which is the reciprocal of insulin sensitivity (%S) (100/%S) as a percentage of a normal reference population (normal young adults). A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean serum insulin concentration two hours post glucose challenge (Oral Glucose Tolerance Test [OGTT]) | Baseline (Day 1) and End of treatment (Day 85)
  Fasting blood samples are taken at 0 minutes prior to a glucose drink and at 30 and 120 minutes post drink. The OGTT measures the serum insulin levels at two hours (120 minutes) compared to 0 minutes. The extent of the elevation in serum insulin levels following a glucose drink are compared between baseline and the end of treatment. An increase in the elevation of serum insulin levels from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean pro-insulin concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of pro-insulin concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean C-peptide concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of C-peptide concentrations. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean beta cell function measured by Homeostasis Model Assessment 2 (HOMA2-%B). | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of beta cell function calculated by HOMA2. HOMA2 is a computer model that uses fasting plasma insulin and glucose concentrations to estimate beta cell function (%B) as a percentage of a normal reference population (normal young adults). An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean Body Mass Index (BMI). | Baseline (Day 1) and End of treatment (Day 85)
  Body Mass Index (kg/m^2) is calculated at baseline and the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean serum total cholesterol concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of serum total cholesterol concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean serum High Density Lipoprotein (HDL)-cholesterol concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of serum HDL-cholesterol. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean serum triglyceride concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for measurement of serum triglyceride concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean C-reactive protein (CRP) concentration. | Baseline (Day 1) and End of treatment (Day 85)
  At baseline and at the end of treatment, a fasting blood sample is taken for high sensitivity measurement of CRP concentrations. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean blood pressure. | Baseline (Day 1) and End of treatment (Day 85)
  Blood pressure is measured at baseline and at the end of treatment. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean Diabetes Treatment Satisfaction Questionnaire (DTSQ): Overall Treatment Satisfaction total score. | Baseline (Day 1) and End of treatment (Day 85)
  The DTSQ (status version) is a self-administered questionnaire consisting of eight items. Six of the eight items are rated from 0 (very dissatisfied, inconvenient, inflexible, etc.) to 6 (very satisfied, convenient, flexible, etc.) and are summed to produce an Overall Treatment Satisfaction score. As such, an increase from baseline to the end of treatment, a positive value, indicates an improvement.
Change from baseline to the end of treatment in mean Diabetes Treatment Satisfaction Questionnaire (DTSQ): Glycaemic Control total score. | Baseline (Day 1) and End of treatment (Day 85)
  The DTSQ (status version) is a self-administered questionnaire consisting of eight items. Two of the eight items are used to assess 'perceived frequency of hyperglycaemia' and 'perceived frequency of hypoglycaemia', both of which are rated from 0 (none of the time) to 6 (most of the time) and are summed to produce a Glycaemic Control score. As such, a decrease from baseline to the end of treatment, a negative value, indicates an improvement.
Change from baseline to the end of treatment in mean overall health Visual Analogue Scale (0-100) total score. | Baseline (Day 1) and End of treatment (Day 85)
  Participants are asked to assess their overall health status using a health Visual Analogue Scale (0-100), where 100 is 'the best health you can imagine' and 0 is 'the worst health you can imagine'. An increase from baseline to the end of treatment, a positive value, indicates an improvement.
Incidence of adverse events (AEs) as a measure of patient safety. | Screening (Day -7) to Final follow-up (Day 92)
  The incidence of treatment-emergent AEs is recorded for the study duration, and the number of participants who experienced an adverse event is presented.
Change from baseline to the end of treatment in mean Beck Depression Inventory-II (BDI-II) total score. | Baseline (Day 1) and End of treatment (Day 85)
  The BDI-II is a multiple choice self-reported inventory that is one of the most widely used instruments for measuring the severity of depression. There are 21 questions or items, each having four possible responses. Each response is assigned a score ranging from zero to three, indicating the severity of the symptom. Items 1 to 13 assess symptoms that are psychological in nature, while items 14 to 21 assess symptoms that are more physical. The sum of all BDI-II item scores indicates the severity of depression. For participants eligible for this study, a score of 21 or over represents depression. The BDI-II can distinguish between different subtypes of depressive disorders, such as major depression and dysthymia. A decrease from baseline to the end of treatment, a negative value, indicates an improvement.
The number of participants with a treatment-emergent flag using the Columbia-Suicide Severity Rating Scale (C-SSRS) during the course of the study. | Baseline (Day 1) to End of treatment (Day 85)
  Participants are scored at each clinic visit for the following outcomes using the C-SSRS: suicidal ideation, suicidal behaviour, suicidality (including complete suicidality). Possible flags are as follows: "Wish to be Dead", "Non-specific Active Suicidal Thoughts", "Active Suicidal Ideation Without Intent", "Active Suicidal Ideation With Intent, No Plan", "Active Suicidal Ideation With Intent and Plan". The number of participants with a treatment-emergent flag is presented.
Incidence of hypoglycaemic episodes during the course of the study. | Screening (Day -7) to End of treatment (Day 85)
  The incidence of treatment-emergent hypoglycaemic episodes (blood glucose concentration below 3 mmol/L) is recorded for the study duration, and the number of participants who experienced a hypoglycaemic episode is presented.
Change from baseline to the end of study in mean Cannabis Withdrawal Scale (CWS) total score. | Baseline (Day 1) and Final follow-up (Day 92)
  The CWS is validated and used as a diagnostic instrument in clinical and research settings where regular monitoring of withdrawal symptoms is required. The CWS will be completed for UK-based participants only. The CWS is a 19 item scale with each item (withdrawal symptom) measured on a 0-10 point scale (0 = Not at all, 5 = moderately, 10 = Extremely). For each item, the participant is asked to record the extent to which it was experienced in the last 24 hours and also to rate its negative impact on their normal daily activities (i.e., two separate scores are recorded for each item using the same 0-10 scale). Scores are summed over the 19 items for each measure, extent of experience and negative impact on normal daily activities. An increase from baseline to the end of study, a positive value, indicates withdrawal.

CONTACTS AND LOCATIONS:
Locations (25):
- Romania (14):
  - Diabol SRL, Brasov
  - Nicodiab SRL, Bucharest
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Institutul National de Diabet, Bucharest
  - Centrul Medical 'Sanatatea Ta' SRL, Bucharest
  - ArtMedical Clinic, Bucharest
  - Societatea Civila Medicala dr. Paveliu, Bucharest
  - Consultmed SRL, Iași
  - Cabinet Medical Individual Diabet Nutritie si Boli Metabolice, Maramures
  - Grandmed SRL, Oradea
  - Spitalul Judetean de Urgente Satu Mare, Satu Mare
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Gagiu D. Remus Cabinet Medical Individual, Târgovişte
  - Mediab SRL Diabet Zaharat, Târgu Mureş
- United Kingdom (11):
  - Avondale Surgery, Chesterfield, Derbyshire
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Aintree University Hospitals NHS Foundation Trust, Liverpool, Merseyside
  - Strensall Medical Practice, York, North Yorkshire
  - Churchill Hospital, Oxford, Oxfordshire
  - Hathaway Surgery, Chippenham, Wiltshire
  - Avenue Surgery, Warminster, Wiltshire
  - St Chad's Surgery, Bath
  - Barts and The London NHS Trust, London